CLINICAL TRIAL: NCT05369533
Title: Dopaminergic Enhancement of Rehabilitation Therapy Early After Stroke
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Steven C. Cramer, MD, FAAN, FAHA, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-000104
Record Dates: First submitted 2022-04-22; First posted 2022-05-11 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: stroke; rehabilitation; telehealth; dopamine
MeSH Terms: conditions — Stroke | interventions — Telerehabilitation; carbidopa, levodopa drug combination

STUDY DESIGN:
Intervention Model Description: Patients are randomized to TR + placebo, TR + Sinemet, or usual care
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded, placebo controlled, randomized. Participants and investigators will be blinded to the study group allocations (placebo vs Sinemet).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Telerehabilitation + Sinemet (Active Comparator): Patients will receive 36 telerehabilitation sessions targeting arm motor function. TR consists of 70 minutes/day of activities targeting arm function, 6 days/week for 6-8 weeks. Half of these sessions are supervised by a licensed therapist, and the other half are done independently. Sinemet is taken one hour before starting TR, for the first 18 sessions.
  Interventions: Device: Telerehabilitation; Drug: Sinemet Pill
- Telerehabilitation + Placebo (Placebo Comparator): Patients will receive 36 telerehabilitation sessions targeting arm motor function. TR consists of 70 minutes/day of activities targeting arm function, 6 days/week for 6-8 weeks. Half of these sessions are supervised by a licensed therapist, and the other half are done independently. Placebo is taken one hour before starting TR, for the first 18 sessions.
  Interventions: Device: Telerehabilitation; Drug: Placebo
- Usual care (No Intervention): Participants in the usual care group will receive no TR or study pill, but will continue with the recommendations made by their care team. All participants will be offered TR at the end of the study.

INTERVENTIONS:
Device: Telerehabilitation — The telerehabilitation system will deliver rehabilitation treatment sessions via a secured internet-connected computer. TR sessions will be a combination of games, exercises, stroke education, assessments, in addition to videoconferencing with therapists to discuss progress, issues, goals, and changes to the treatment plan.
  Arms: Telerehabilitation + Placebo; Telerehabilitation + Sinemet
Drug: Sinemet Pill — Sinemet 25/100 will be taken 1 hour prior to TR, for the first 18 sessions.
  Arms: Telerehabilitation + Sinemet
Drug: Placebo — Placebo will be taken 1 hour prior to TR, for the first 18 sessions.
  Arms: Telerehabilitation + Placebo

SUMMARY:
This study explores the effects of telerehabilitation and a study medication on rehabilitation outcomes in patients with stroke resulting in arm weakness. Patients with arm weakness due to a stroke that happened in the past 30 days will be randomized into one of three groups: [1] TR and placebo (a sugar pill) on top of usual care; [2] TR and a medication (Sinemet 25/100) on top of usual care; [3] or usual care alone (no TR and no pill, but people in this group will be offered TR once the study is done). TR consists of 70 minutes/day of activities targeting arm function, 6 days a week for 6 weeks.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study that involves the use of telerehabilitation to deliver additional therapy for persons with stroke. Participants with arm weakness due to a stroke in the past 30 days will be randomized into one of three groups: (1) TR + Sinemet on top of usual care, (2) TR + placebo (sugar pill) on top of usual care, or (3) usual care only (no TR, no pill). The hypothesis of this study is patients receiving TR will have significantly greater recovery of arm function compared to patients receiving usual care. In addition, Sinemet is hypothesized to significantly enhancing this improvement.

Study participation will last up to 3 months and includes 4 in-person visits. At these visits, patients will undergo a battery of assessments including arm function, a single MRI scan of the brain, and blood draw for genotyping. Patients undergoing TR will receive arm motor training, which consists of 36 sessions of of assigned exercises, games, and stroke education; these are 70 minutes in length and take 6 days a week over 6-8 weeks. Subjects receiving TR will take a pill (Sinemet or placebo) prior to the TR training for the first 18 TR sessions; TR subjects will also continue usual care. Patients in the usual care group will not engage in TR or take a study pill, but will instead continue all of the therapies recommended by their medical team. At the end of the study, participants in the usual care group will be offered TR.

ELIGIBILITY:
INCLUSION CRITERIA

1. Age 18 years or older
2. Stroke that has been radiologically verified and has time of onset 30 days or less from the time of randomization
3. ARAT score of <32 (out of 57) at Visit 1
4. At Visit 1, either

   1. BBT score with affected arm is at least 1 block in 60 seconds OR
   2. There is a visible flicker in each of the following movements with gravity eliminated: wrist extension and finger flexion
5. At Visit 1, either

   1. The range of motion against gravity must be ≥45 degrees in both the paretic shoulder and elbow OR
   2. the patient must be able to use at least 3 different telerehab system input devices
6. Informed consent and behavioral contract signed by the subject (i.e., no surrogate consent)

EXCLUSION CRITERIA

1. A major, active, coexistent neurological or psychiatric disease (e.g., alcoholism or dementia)
2. Major medical disorder that reduces subject's ability to comply with study procedures
3. Severe depression, defined as CES-D score >24 at screening visit
4. Significant cognitive impairment, defined as presence of either

   1. Montreal Cognitive Assessment (MoCA) score <22 OR
   2. Trail Making Test: Part A score ≤14
   3. Note that lower scores may be permitted if due to aphasia and if the patient is specifically allowed by Dr. Cramer
5. Deficits in communication that interfere with reasonable study participation
6. Lacking visual acuity, with or without corrective lens, of 20/50 or better in at least one eye
7. Life expectancy <6 months
8. Pregnant
9. Botox to arms, legs or trunk in the preceding 4 months, or expectation that Botox will be administered to the arm, leg or trunk within 3 months of study enrollment
10. Unable to successfully perform all 3 rehabilitation exercise test examples
11. Unable or unwilling to perform study procedures/therapy or attend study visits, or expectation of noncompliance with study procedures/therapy
12. Non-English or non-Spanish speaking, such that subject does not speak either language sufficiently to comply with study procedures
13. Isolation due to active COVID-19
14. Any contraindication to L-Dopa:

    1. Patient is currently taking a monoamine oxidase inhibitor; if the patient took such a drug in the past, it must be discontinued at least two weeks prior to study enrollment
    2. Known hypersensitivity to any component of Sinemet
    3. Narrow-angle glaucoma; if wide-angle glaucoma is present, the patient can only be enrolled with explicit written approval from their ophthalmologist
    4. History of melanoma or suspected melanoma
    5. Patient is currently taking phenytoin, papaverine, isoniazid, or a dopamine D2 receptor antagonist (such as a phenothiazine, butyrophenone, or risperidone)
    6. Currently taking a direct dopaminergic agonist
15. Expectation that subject will not have single domicile address during 6 weeks of therapy that has either Verizon wireless reception or a home WiFi network and that has space for TR system, and is within 30 miles of Cal Rehab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Cramer, Principal Investigator — University of California, Los Angeles
Locations (1):
- California Rehabilitation Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset will be shared with appropriate personnel after the main study manuscript is published
Supporting Information: Study Protocol, SAP
Time Frame: likely starting 1-2 years after study completion, lasting for several years thereafter
Access Criteria: Data will be shared using common data formats with appropriate personnel

REFERENCES:
- [Background] Dodakian L, McKenzie AL, Le V, See J, Pearson-Fuhrhop K, Burke Quinlan E, Zhou RJ, Augsberger R, Tran XA, Friedman N, Reinkensmeyer DJ, Cramer SC. A Home-Based Telerehabilitation Program for Patients With Stroke. Neurorehabil Neural Repair. 2017 Oct-Nov;31(10-11):923-933. doi: 10.1177/1545968317733818. Epub 2017 Oct 26. PMID 29072556
- [Background] Chen Y, Abel KT, Janecek JT, Chen Y, Zheng K, Cramer SC. Home-based technologies for stroke rehabilitation: A systematic review. Int J Med Inform. 2019 Mar;123:11-22. doi: 10.1016/j.ijmedinf.2018.12.001. Epub 2018 Dec 11. PMID 30654899
- [Background] Cramer SC, Dodakian L, Le V, See J, Augsburger R, McKenzie A, Zhou RJ, Chiu NL, Heckhausen J, Cassidy JM, Scacchi W, Smith MT, Barrett AM, Knutson J, Edwards D, Putrino D, Agrawal K, Ngo K, Roth EJ, Tirschwell DL, Woodbury ML, Zafonte R, Zhao W, Spilker J, Wolf SL, Broderick JP, Janis S; National Institutes of Health StrokeNet Telerehab Investigators. Efficacy of Home-Based Telerehabilitation vs In-Clinic Therapy for Adults After Stroke: A Randomized Clinical Trial. JAMA Neurol. 2019 Sep 1;76(9):1079-1087. doi: 10.1001/jamaneurol.2019.1604. PMID 31233135
- [Background] Chen Y, Chen Y, Zheng K, Dodakian L, See J, Zhou R, Chiu N, Augsburger R, McKenzie A, Cramer SC. A qualitative study on user acceptance of a home-based stroke telerehabilitation system. Top Stroke Rehabil. 2020 Mar;27(2):81-92. doi: 10.1080/10749357.2019.1683792. Epub 2019 Nov 4. PMID 31682789
- [Background] Cramer SC, Dodakian L, Le V, McKenzie A, See J, Augsburger R, Zhou RJ, Raefsky SM, Nguyen T, Vanderschelden B, Wong G, Bandak D, Nazarzai L, Dhand A, Scacchi W, Heckhausen J. A Feasibility Study of Expanded Home-Based Telerehabilitation After Stroke. Front Neurol. 2021 Feb 3;11:611453. doi: 10.3389/fneur.2020.611453. eCollection 2020. PMID 33613417
- [Background] Paik SM, Cramer SC. Predicting motor gains with home-based telerehabilitation after stroke. J Telemed Telecare. 2023 Dec;29(10):799-807. doi: 10.1177/1357633X211023353. Epub 2021 Jun 22. PMID 34156873
- [Background] Pearson-Fuhrhop KM, Cramer SC. Pharmacogenetics of neural injury recovery. Pharmacogenomics. 2013 Oct;14(13):1635-43. doi: 10.2217/pgs.13.152. PMID 24088134

RESULTS

PARTICIPANT FLOW:
Groups:
- Telerehabilitation + Sinemet: Patients will receive 36 telerehabilitation (TR) sessions targeting arm motor function. TR consists of 70 minutes/day of activities targeting arm function, 6 days/week for 6-8 weeks. Half of these sessions are supervised by a licensed therapist, and the other half are done independently. A study pill (Sinemet) is taken one hour before starting TR, for the first 18 sessions.
  Telerehabilitation: The telerehabilitation system will deliver rehabilitation treatment sessions via a secured internet-connected computer. TR sessions will be a combination of games, exercises, stroke education, assessments, in addition to videoconferencing with therapists to discuss progress, issues, goals, and changes to the treatment plan.
- Telerehabilitation + Placebo: Patients will receive 36 telerehabilitation (TR) sessions targeting arm motor function. TR consists of 70 minutes/day of activities targeting arm function, 6 days/week for 6-8 weeks. Half of these sessions are supervised by a licensed therapist, and the other half are done independently. A study pill (placebo) is taken one hour before starting TR, for the first 18 sessions.
  Telerehabilitation: The telerehabilitation system will deliver rehabilitation treatment sessions via a secured internet-connected computer. TR sessions will be a combination of games, exercises, stroke education, assessments, in addition to videoconferencing with therapists to discuss progress, issues, goals, and changes to the treatment plan.
Period: Overall Study
Arm/Group | Telerehabilitation + Sinemet | Telerehabilitation + Placebo | Usual Care
Started | 6 | 10 | 9
Completed | 4 | 8 | 9
Not Completed | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Telerehabilitation + Sinemet: Patients will receive 36 telerehabilitation sessions targeting arm motor function. TR consists of 70 minutes/day of activities targeting arm function, 6 days/week for 6-8 weeks. Half of these sessions are supervised by a licensed therapist, and the other half are done independently. A study pill (Sinemet) is taken one hour before starting TR, for the first 18 sessions.
  Telerehabilitation: The telerehabilitation system will deliver rehabilitation treatment sessions via a secured internet-connected computer. TR sessions will be a combination of games, exercises, stroke education, assessments, in addition to videoconferencing with therapists to discuss progress, issues, goals, and changes to the treatment plan.
- Telerehabilitation + Placebo: Patients will receive 36 telerehabilitation sessions targeting arm motor function. TR consists of 70 minutes/day of activities targeting arm function, 6 days/week for 6-8 weeks. Half of these sessions are supervised by a licensed therapist, and the other half are done independently. A study pill (Placebo) is taken one hour before starting TR, for the first 18 sessions.
- Total: Total of all reporting groups
Arm/Group | Telerehabilitation + Sinemet | Telerehabilitation + Placebo | Usual Care | Total
Number analyzed (Participants) | 6 | 10 | 9 | 25
Age, Continuous [Mean (Full Range); unit: years] | 59.8 [33 to 80] | 65.2 [45 to 92] | 66.4 [54 to 82] | 64.4 [33 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 3 | 8
  Male | 6 | 5 | 6 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Black or African American | 2 | 3 | 1 | 6
  White | 2 | 5 | 7 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Action Research Arm Test [Mean (Standard Deviation); unit: units on a scale] | 20.7 (8.9) | 18 (12.2) | 18.3 (12.7) | 18.8 (11.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Action Research Arm Test Score From Baseline to 3 Months
Description: Measures arm function using a scale that runs from 0 to 57 points, with higher scores indicating greater arm function.
Time Frame: Measured at baseline and 3 months later
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Telerehabilitation + Sinemet: Patients will receive 36 telerehabilitation sessions targeting arm motor function. TR consists of 70 minutes/day of activities targeting arm function, 6 days/week for 6-8 weeks. Half of these sessions are supervised by a licensed therapist, and the other half are done independently. Patients will take Sinemet one hour before starting TR, for the first 18 sessions.
  Telerehabilitation: The telerehabilitation system will deliver rehabilitation treatment sessions via a secured internet-connected computer. TR sessions will be a combination of games, exercises, stroke education, assessments, in addition to videoconferencing with therapists to discuss progress, issues, goals, and changes to the treatment plan.
  Sinemet Pill: Sinemet 25/100 will be taken 1 hour prior to TR, for the first 18 sessions.
- Telerehabilitation + Placebo: Patients will receive 36 telerehabilitation sessions targeting arm motor function. TR consists of 70 minutes/day of activities targeting arm function, 6 days/week for 6-8 weeks. Half of these sessions are supervised by a licensed therapist, and the other half are done independently. Patients will take a study pill (placebo) one hour before starting TR, for the first 18 sessions.
  Telerehabilitation: The telerehabilitation system will deliver rehabilitation treatment sessions via a secured internet-connected computer. TR sessions will be a combination of games, exercises, stroke education, assessments, in addition to videoconferencing with therapists to discuss progress, issues, goals, and changes to the treatment plan.
Arm/Group | Telerehabilitation + Sinemet | Telerehabilitation + Placebo | Usual Care
Number analyzed (Participants) | 6 | 10 | 9
score on a scale | 23.5 (6.8) | 24 (13.7) | 15.1 (7.8)

2. Secondary Outcome: Change in Arm Motor Fugl-Meyer Scale From Baseline to 3 Months
Description: Measures arm motor impairment using a scale that runs from 0 to 66 points, with higher scores indicating greater arm motor function (less impairment)
Time Frame: Measured at baseline and 3 months later
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telerehabilitation + Sinemet | Telerehabilitation + Placebo | Usual Care
Number analyzed (Participants) | 6 | 10 | 9
score on a scale | 23.8 (5.4) | 21.9 (12) | 12 (5.6)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Telerehabilitation + Sinemet | Telerehabilitation + Placebo | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/6 | 3/10 | 4/9
Other Adverse Events (participants affected / at risk) | 2/6 | 1/10 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telerehabilitation + Sinemet (N=6) | Telerehabilitation + Placebo (N=10) | Usual Care (N=9)
Hospitalization (unrelated to study procedures) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) — Fall
Hospitalization due to GI-related issues (unrelated to study procedures) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hospitalization due to fluid build-up (unrelated to study procedures) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) — Pleural effusion, pulmonary edema
Hospitalization due to cardiac issues (unrelated to study procedures) (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hospitalization due to neurological issue (unrelated to study procedures) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telerehabilitation + Sinemet (N=6) | Telerehabilitation + Placebo (N=10) | Usual Care (N=9)
Loss of balance (unrelated to study) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pain (not related to study) (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT05369533/Prot_SAP_000.pdf